CLINICAL TRIAL: NCT06103877
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of AZD1163 Administered as Single and Multiple Ascending Doses in Healthy Volunteers
Brief Title: A Placebo-controlled Safety and Tolerability Study of Intravenous (IV) and Subcutaneous (SC) AZD1163 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D9640C00001
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Rheumatoid arthritis; Pharmocokinetics; Healthy volunteers
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (20):
- Part 1 Cohort 1 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 2 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 3 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 4 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 5a SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 5b SAD (Active Comparator): Participants will receive SC injection of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 6 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 7 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Cohort 8 SAD (Active Comparator): Participants will receive IV infusion of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Pooled Placebo SAD IV (Placebo Comparator): Participants will receive matching IV infusion of placebo on Day 1.
  Interventions: Other: Placebo
- Part 1 Placebo SAD SC (Placebo Comparator): Participants will receive matching SC injection of placebo on Day 1.
  Interventions: Other: Placebo
- Part 1 Cohort 9 SAD (Chinese Participants) (Active Comparator): Participants will receive SC injection of AZD1163 on Day 1.
  Interventions: Biological: AZD1163
- Part 1 Placebo SAD (Chinese Participants) (Placebo Comparator): Participants will receive matching SC injection of placebo on Day 1.
  Interventions: Other: Placebo
- Part 2 Cohort 1 MAD (Global) (Active Comparator): Participants will receive SC injection of AZD1163 on Days 1 and 15.
  Interventions: Biological: AZD1163
- Part 2 Cohort 2 MAD (Global) (Active Comparator): Participants will receive SC injection of AZD1163 on Days 1 and 15.
  Interventions: Biological: AZD1163
- Part 2 Placebo MAD (Global) (Placebo Comparator): Participants will receive matching SC injection of placebo on Days 1 and 15.
  Interventions: Other: Placebo
- Part 2 Cohort 3 MAD (Chinese Participants) (Active Comparator): Participants will receive SC injection of AZD1163 on Days 1 and 15.
  Interventions: Biological: AZD1163
- Part 2 Cohort 4 MAD (Japanese participants) (Active Comparator): Participants will receive SC injection of AZD1163 on Days 1 and 15.
  Interventions: Biological: AZD1163
- Part 2 Placebo MAD (Chinese participants) (Placebo Comparator): Participants will receive matching SC injection of placebo on Days 1 and 15.
  Interventions: Other: Placebo
- Part 2 Placebo MAD (Japanese participants) (Placebo Comparator): Participants will receive matching SC injection of placebo on Days 1 and 15.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AZD1163 — In Part 1, Participants will receive AZD1163 through IV infusion or SC injection on Day 1.
  In Part 2, participants will receive AZD1163 through SC injection on Days 1 and 15.
  Arms: Part 1 Cohort 1 SAD; Part 1 Cohort 2 SAD; Part 1 Cohort 3 SAD; Part 1 Cohort 4 SAD; Part 1 Cohort 5a SAD; Part 1 Cohort 5b SAD; Part 1 Cohort 6 SAD; Part 1 Cohort 7 SAD; Part 1 Cohort 8 SAD; Part 1 Cohort 9 SAD (Chinese Participants); Part 2 Cohort 1 MAD (Global); Part 2 Cohort 2 MAD (Global); Part 2 Cohort 3 MAD (Chinese Participants); Part 2 Cohort 4 MAD (Japanese participants)
Other: Placebo — In Part 1, Participants will receive matching placebo through IV infusion or SC injection on Day 1.
  In Part 2, participants will receive matching placebo through SC injection on Days 1 and 15.
  Arms: Part 1 Placebo SAD (Chinese Participants); Part 1 Placebo SAD SC; Part 1 Pooled Placebo SAD IV; Part 2 Placebo MAD (Chinese participants); Part 2 Placebo MAD (Global); Part 2 Placebo MAD (Japanese participants)

SUMMARY:
A study to demonstrate the safety and tolerability of AZD1163 when administered intravenously and subcutaneously in healthy participants.

DETAILED DESCRIPTION:
This is a first time in human (FTiH), placebo-controlled, sequential study in healthy participants. This study consists of two parts: Part 1 Single Ascending Dose (SAD) and Part 2 Multiple Ascending Dose (MAD). Part 1 will contain 9 cohorts, 8 intravenously (IV) administered dose levels and 1 subcutaneously (SC) administered dose level of AZD1163. Part 2 will contain 2 SC dose levels of AZD1163. A sentinel dosing approach will be taken. Each participant will be involved in the study for approximately 70 weeks.

The study will comprise of:

* A Screening Period of maximum 28 days for both Part 1 and Part 2.
* Part 1: A single dose of AZD1163 with an in-clinic period of 7 to 8 days.
* Part 2: Two doses of AZD1163, given 2 weeks apart both with an in-clinic period of 7 to 8 days.
* An outpatient Follow-up Period of approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants with suitable veins for cannulation or repeated venipuncture
* All females must have a negative pregnancy test
* Females of childbearing potential must not be lactating and, if heterosexually active, agree to taking approved method/s of contraception
* BMI between 18 and 32 kg/m^2 and weigh at least 45 kg

Exclusion Criteria:

* Has received another new chemical entity
* History of any disease or disorder which may put participant at risk in the study
* Current or recurrent disease of clinical significance
* Medical history of malignancies except for cervical carcinoma and non-melanoma skin cancer (NMSC)
* Any clinically important illness, medical/procedure, or trauma
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis result at screening
* Any positive result on screening for serum hepatitis B surface antigen (HbsAg), hepatitis B core antibody (HbcAb), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV)
* History of latent or active tuberculosis (TB) or exposure to endemic areas
* Evidence of active TB or untreated/inadequately/inappropriately treated for latent TB
* Positive testing for Covid-19 prior to dosing, case of Covid-19 within 4 weeks, or long-term Covid-19-related sequelae
* Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing or presence of fever
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead electrocardiogram (ECG), and any clinically important abnormalities in the 12-lead ECG
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From Day -1 until end of study (Day 450)
  To assess the safety and tolerability of single and multiple ascending doses of AZD1163 following IV or SC administration.

SECONDARY OUTCOMES:
Area under plasma concentration-time curve from zero extrapolated to infinity (AUCinf) | Part 1: Days 1-8, 11, 15, 22, 29, 57, 113, 225, 281, 365, 450; Part 2: Days 1-8, 11, 15-16, 22, 29, 57, 113, 225, 281, 365, 450
  To characterize the pharmacokinetics (PK) of AZD1163 following IV/SC administration of single and multiple ascending doses.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Part 1: Days 1-8, 11, 15, 22, 29, 57, 113, 225, 281, 365, 450; Part 2: Days 1-8, 11, 15-16, 22, 29, 57, 113, 225, 281, 365, 450
  To characterize the PK of AZD1163 following IV/SC administration of single and multiple ascending doses.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Part 1: Days 1-8, 11, 15, 22, 29, 57, 113, 225, 281, 365, 450; Part 2: Days 1-8, 11, 15-16, 22, 29, 57, 113, 225, 281, 365, 450
  To characterize the PK of AZD1163 following SC administration of single and multiple ascending doses.
Volume of distribution (apparent) at steady state following extravascular administration (Vz/F) | Part 1: Days 1-8, 11, 15, 22, 29, 57, 113, 225, 281, 365, 450; Part 2: Days 1-8, 11, 15-16, 22, 29, 57, 113, 225, 281, 365, 450
  To characterize the PK of AZD1163 following SC administration of single and multiple ascending doses.
Maximum observed plasma (peak) drug concentration (Cmax) | Part 1: Days 1-8, 11, 15, 22, 29, 57, 113, 225, 281, 365, 450; Part 2: Days 1-8, 11, 15-16, 22, 29, 57, 113, 225, 281, 365, 450
  To characterize the PK of AZD1163 following IV/SC administration of single and multiple ascending doses.
Number of participants with positive anti-AZD1163 antibodies | Part 1: Day 1, 11, 29, 113, 225, 281, 365, 450; Part 2: Day 1, 15, 29, 57, 113, 281, 365, 450
  To evaluate the immunogenicity of AZD1163.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/